CLINICAL TRIAL: NCT00948454
Title: The Dose Effect Of Cigarette-Smoking On Indices Of Arterial Function And Oxidative Stress
Brief Title: Research Study on the Effects of Smoking on Arteries
Status: Completed | Type: Observational
Sponsor: University of Pennsylvania (Other)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: Garret A. FitzGerald Chair Department of Pharmacology Director, Institute for Translational Medicine & Therapeutics, University of Pennsylvania
Other Study IDs: 704074; 0775
Record Dates: First submitted 2009-07-28; First posted 2009-07-29 (Estimated); Last update posted 2009-10-27 (Estimated); Status verified 2009-10

CONDITIONS: Smoking
Keywords: smoking
MeSH Terms: conditions — Smoking

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Buffy coat from 4ml of blood will be stored for future genomic and proteomic analysis. Blood will also be collected for telemore length. This will be performed at an outside institution. Identifiers will be stripped from the samples prior to send out.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Light smokers: 2 blood draws, 3 urine collections and a test called an FMD which tests the circulation in your arm via ultrasound will be performed on the study day. Subjects will bring their own cigarettes on that day and smoke their regular amount. Female subjects will also have a pregnancy test done on the test day.
- Heavy Smokers: 2 blood draws, 3 urine collections and a test called an FMD which tests the circulation in your arm via ultrasound will be performed on the study day. Subjects will bring their own cigarettes on that day and smoke their regular amount. Female subjects will also have a pregnancy test done on the test day.
- Non Smokers: 2 blood draws, 3 urine collections and a test called an FMD which tests the circulation in your arm via ultrasound will be performed on the study day. Female subjects will also have a pregnancy test done on the test day.

SUMMARY:
The current proposal, will elucidate the role of oxidant stress (OS) on arterial function as measured by flow mediated vasodilation. In addition, the investigators will address the hypothesis, that a pro-oxidant might have different degrees of effects on different biological targets, by performing quantitative assessment of the effects of OS on lipids, proteins and DNA.

ELIGIBILITY:
Inclusion Criteria:

* Chronic smokers (of between 4 and 20 years duration) and non-smokers will be recruited to the GCRC. Smokers will be allocated to a "light" group, smoking 4-10 cigarettes per day and a "heavy" smoking group who smoke 11-20 cigarettes per day.
* Non-smokers will be defined as those with a life time consumption of no more than 20 cigarettes, do not live or work in a smoky atmosphere.
* All individuals will have a normal history and clinical examination, including a normal EKG, urinalysis and serum chemistry, haemogram and negative urinary pregnancy test.

Exclusion Criteria:

* previously suffered an acute major cardiovascular event
* those with a chronic disease
* those taking chronic medication
* those with a history of alcoholism or substance abuse
* Ex-smokers
* Subjects, who have less than or equal to 60% platelet aggregation in response to arachidonic acid

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Chronic smokers (of between 4 and 20 years duration) and non-smokers will be recruited. Smokers will be allocated to a "light" group, smoking 4-10 cigarettes per day and a "heavy" smoking group who smoke 11-20 cigarettes per day. Non-smokers will be defined as those with a life time consumption of no more than 20 cigarettes, do not live or work in a smoky atmosphere. All individuals will have a normal history and clinical examination, including a normal EKG, urinalysis and serum chemistry, haemogram and negative urinary pregnancy test.
Sampling Method: Non-Probability Sample
Enrollment: 105 (Actual)
Dates: Start 2003-01; Primary Completion 2006-05 (Actual); Study Completion 2006-06 (Actual)

PRIMARY OUTCOMES:
To assess the dose-related effects of cigarette smoking on flow mediated arterial function in humans. | Study Day

SECONDARY OUTCOMES:
To assess the dose-related effects of cigarette smoking on COX activation. | Twice during study day
To assess the dose-related effects of cigarette smoking on novel indices of lipid peroxidation, protein oxidation and DNA modification by lipid adducts. | Study day

CONTACTS AND LOCATIONS:
Overall Officials: Garret A FitzGerald, MD, Principal Investigator — University of Pennsylvania
Locations (1):
- University of Pennsylvania, Philadelphia, Pennsylvania, United States